CLINICAL TRIAL: NCT06827743
Title: Effectiveness of Feeding Intervention on Feeding Behavior, Developmental Areass and Sensory Processing in Children with Cerebral Visual Impairment and Cerebral Palsy: a Pilot Randomized Controlled Trial
Brief Title: Feeding Behavior Intervention in Children with Cerebral Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, mustafa cemali, Assist. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/186
Record Dates: First submitted 2025-02-08; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Feeding Behavior; Sensory Integration Disorder; Cerebral Visual Impairment
Keywords: Feeding Behavior; Sensory Integration Disorder; Cerebral Visual Impairment; Cerebral palsy
MeSH Terms: conditions — Feeding Behavior; Blindness, Cortical; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled intervention trial
Who Masked: Investigator
Masking Description: The clinician who conducted the assessment and the clinician who implemented the intervention were different individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral visual impairment intervention group (Experimental): In addition to sensory integration training, nutritional behavior training will be given to this group.
  Interventions: Behavioral: feeding behavior education; Behavioral: Sensory integration intervention
- Ceerbral visual impairment children (control group) (Active Comparator): Only sensory integration training will be given to this group.
  Interventions: Behavioral: Sensory integration intervention

INTERVENTIONS:
Behavioral: feeding behavior education — Two groups will receive personalized sensory integration training, and one group will receive feeding behavior training. Both the caregiver and the child will take part in feeding behavior training. In order for the training to be successful, the therapist, child, and parent cooperation is necessary. Before this training, the children will be evaluated with the Behavioral Pediatric Feeding Assessment Scale and a behavioral training plan will be created according to the children's attitudes and behaviors during feeding. This plan will include organizing feeding times, determining the family's approach to the child's behaviors during feeding, regulating the children's feeding behavior problems with extinguishing and desensitization methods, and organizing the feeding environment, and creating a personalized training plan.
  Arms: Cerebral visual impairment intervention group
Behavioral: Sensory integration intervention — The sensory integration training given to both groups includes training that includes oral processing skills in particular, as well as training that includes tactile, vestibular, proprioception, and visual stimuli as needed. Children will be supported with sensory stimuli in order to ensure that the child focuses and remains calm. Sensory integration training will be planned by taking into account the Dunn Sensory Profile test results. In this training, different patterned fabrics, plushes, and toys with different surfaces for tactile stimulation will be provided to maintain the child's calmness and focus; swings and exercise balls for vestibular stimulation; and training to provide sensory regulation with proprioceptive approaches. In addition, within the scope of sensory integration training, stimuli will be provided in the oral region according to the children's sensory responses to the texture, taste, and content of foods.

SUMMARY:
This study was planned to investigate the effects of nutritional education given in addition to sensory integration intervention on feeding behavior, sensory processing and developmental areas in children with Cerebral Visual Impairment (CVI) and Cerebral Palsy (CP). Children with CVI and CP were randomly divided into two groups. Sensory integration education was applied to both groups and additional feeding behavior education was applied to one group. The development in feeding behavior and sensory processing was analyzed before and after the intervention.

DETAILED DESCRIPTION:
This study was planned to investigate the effects of feeding education given in addition to sensory integration intervention on feeding behavior, sensory processing and developmental areas in children with CVI and CP. Children with CVI and CP aged 46-60 months were randomly divided into two groups. Sensory integration training was applied to both groups and additional feeding behavior training was applied to 1 group. Before and after the intervention, children's feeding behavior was evaluated with the Behavioral Pediatric Feeding Assessment Scale and sensory processing skills with the Dunn Sensory Profile. The interventions were applied 3 days a week for 12 weeks. Intervention details are as follows.

The duration and protocol of the training were designed by referring to previous studies. The training program includes sensory integration and feeding behavior training. Both the control and study groups will receive 2 sessions of sensory integration-based feeding training of 40 minutes per week for 12 weeks. The study group will receive 2 sessions of feeding behavior training of 40 minutes per week in addition to sensory integration training for 12 weeks. The sensory integration training given to both groups includes training that includes oral processing skills in particular, as well as training that includes tactile, vestibular, proprioception and visual stimuli when needed. The child will be supported with sensory stimuli to ensure that they focus and remain calm. Sensory integration training will be planned considering the Dunn Sensory Profile test results. In this training, different patterned fabrics, plush and toys with different surfaces for tactile stimulation to ensure the child's calmness and focus; swings and exercise balls for vestibular stimulation; and training to provide sensory regulation with proprioceptive approaches will be provided. In addition, within the scope of sensory integration training, stimuli will be given to the oral region according to the children's sensory responses to the texture, taste and content of foods. In addition, oral sensory integration training will be given with sensory stimuli for chewing problems. Two groups will receive personalized sensory integration training, while one group will receive feeding behavior training. Both the caregiver and the child will participate in the feeding behavior training. In order for the training to be successful, the therapist, the child and the parent must cooperate. Before this training, children will be evaluated with the Behavioral Pediatric Feeding Assessment Scale and a behavioral training plan will be created according to the children's attitudes and behaviors during feeding. This plan will include organizing feeding times, determining the families' approach to the child's behavior during feeding, organizing the children's feeding behavior problems with extinguishing and desensitization methods, and organizing the feeding environment. The sensory integration training room was designed according to Parham's sensory integration therapy principles. An individualized sensory integration training based on the basic principles of sensory integration therapy developed by Parham will be applied. According to the evaluations in the individualized program, the baby's problem areas are determined and training is planned in line with certain principles regarding the problem areas. These principles are as follows: Providing sensory opportunities, revealing problem areas, avoiding negative experiences, cooperating in activity choices, helping self-organization, supporting with optimum stimuli, creating a play environment, maximizing the child's success, ensuring physical safety and organizing the child's life within the play environment and ensuring alliance during treatment. All training will be delivered individually, face to face, in therapy rooms in accordance with the sensory integration room plan.

ELIGIBILITY:
Inclusion Criteria:

* • Children with Cerebral Palsy Diagnosed with Cerebral Visual Impairment in Hospital Report

  * Between the ages of 48-72,
  * Having been diagnosed with cerebral palsy.
  * Having a feeding problem according to the results of the behavioral pediatric feeding assessment scale
  * Individuals who volunteer to participate in the study and read and signed the informed consent form by their parents will be included in the study.

Exclusion Criteria:

* Not accepting to participate in the study.

  * Not having any serious sensory loss other than vision problems. (According to the hospital report)
  * Having had any surgery in the last 6 months.
  * Having had very frequent epileptic seizures

Ages: 48 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Behavioral Pediatric Feeding Assessment Scale | 12 weeks
  The Behavioral Pediatric Feeding Assessment Scale, developed by Crist and colleagues, is a 5-point Likert-type scale. The statements in the scale consisting of 25 questions are scored between 1 and 5 (1=Never, 2=Rarely, 3=Sometimes, 4=Frequently, 5=Always). The scores to be obtained from the scale vary between 35-175, and an increase in the obtained score indicates a highly problematic eating disorder and eating habits. The scale consists of four sub-dimensions. There are 7 items in the food selectivity sub-dimension, 5 items in the early food refusal sub-dimension, 5 items in the early lumpy food refusal sub-dimension, and 7 items in the late food refusal sub-dimension. A total score above 84 on the scale or more than 9 problems indicates an eating behavior problem. The Turkish validity and reliability study of the scale was conducted by Önal and colleagues. Cronbach's α value was found to be 0.88.

SECONDARY OUTCOMES:
Dunn Sensory Profile | 12 weeks
  The Sensory Profile developed by Dunn is a 125-question questionnaire used in sensory assessment in children aged 3-10. This questionnaire is answered by the caregiver who is in frequent contact with the child in daily life. It includes questions about many senses such as auditory processing, visual processing, vestibular processing, tactile processing, multi-sensory processing and oral sensory processing. The items are evaluated using 5-point frequency responses between always and never. A higher score for each subdomain means worse sensory processing. The Turkish validity and reliability studies of the scale were conducted by Kayıhan et al. The Cronbach α values of the questionnaire are between 0.63 and 0.97 for all subdomains.

CONTACTS AND LOCATIONS:
Locations (1):
- Special Education Center, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be shared.

REFERENCES:
- [Background] Erol, N., N. Sezgin, and I. Savaşır, Validity studies on Ankara Development Screening Inventory. Turkish Journal of Psychology, 1993. 29(8): p. 16-22.
- [Background] Onal, S., E.Ç. Var, and A. Uçar, Adaptation study of the Behavioral Pediatric Feeding Assessment Scale (BPFAS) to Turkish. Nevşehir Science and Technology Journal, 2017. 6(1): p. 93-101.
- [Background] Kayihan H, Akel BS, Salar S, Huri M, Karahan S, Turker D, Korkem D. DEVELOPMENT OF A TURKISH VERSION OF THE SENSORY PROFILE: TRANSLATION, CROSS-CULTURAL ADAPTATION, AND PSYCHOMETRIC VALIDATION. Percept Mot Skills. 2015 Jun;120(3):971-86. doi: 10.2466/08.27.PMS.120v17x8. Epub 2015 Jun 9. PMID 26057421
- [Background] Dunn, W., Sensory profile. PsycTESTS Dataset, 1999.
- [Background] Lehman, S.S., Cortical Visual Impairment in the Child with Cerebral Palsy. Cerebral Palsy, 2020: p. 1049-1055.